CLINICAL TRIAL: NCT06338072
Title: Impact of the Menstrual Cycle on the Control of Type 1 Diabetes in Reproductive Aged Women Using an Advanced Closed Loop System.
Brief Title: Impact of the Menstrual Cycle in Reproductive Aged Women With Type 1 Diabetes Using a Closed Loop System (DIABETEXX/1).
Acronym: DIABETEXX/1
Status: Recruiting | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Universitat Politècnica de València (Other)
Responsible Party: Sponsor
Other Study IDs: DIABETEXX/1
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes, close loop system, women
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adult women of childbearing age using a loop system.: Adult women of childbearing age using the Minimed 780G loop system. Sixty-nine women of reproductive age will be recruited to assess variations in glycemic control across different stages of the menstrual cycle. Additionally, a subset of these women (n = 50) will wear a wearable device to collect temperature, photoplethysmography, and accelerometry data.
- Adult men under 50 years old using a closed loop system.: A control group of 50 men will wear a wearable device to collect temperature, photoplethysmography, and accelerometry data.

SUMMARY:
The aim of this observational study is to assess the effectiveness of automatic insulin infusion in responding to changes in insulin sensitivity throughout various phases of the menstrual cycle in a cohort of reproductive-aged women with type 1 diabetes, using an advanced closed-loop system. By gaining insights into both the limitations and effectiveness of this adaptation, we aim to inform the enhancement of control algorithms and learning strategies within closed-loop systems. This research is especially vital for addressing the distinct challenges that women commonly encounter in maintaining glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for DM1 according to ADA
* Women and men treated with the Medtronic© MinimedTM 780G advanced closed loop system.
* Women presenting spontaneous regular menstrual cycles with a duration of 24 to 35 days, during the last year.
* Men under 50 years old.
* Acceptance of participation in the study and signing of the informed consent

Exclusion Criteria:

* Gestation
* Use of hormonal contraceptives (including intrauterine devices)
* Institutionalization, serious or terminal illness or renal replacement therapy.
* Refusal to participate in the study or to sign the informed consent

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Gender Based: Yes — Sixty-nine women of reproductive age will be recluted to investigate fluctuations in glycemic control throughout the menstrual cycle. Furthermore, a subgroup comprising 50 of these women, along with a control group consisting of 50 men, will wear a wearable device to gather temperature, photoplethysmography, and accelerometry data
Study Population: Patients of both genders, aged 18 or older, with type 1 diabetes and in their reproductive years, receiving care at the Endocrinology and Nutrition Department of Ramón y Cajal University Hospital in Madrid, and undergoing treatment with the Medtronic© MinimedTM 780G closed loop advanced system.
Sampling Method: Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Time in range | 1 month
  To assess the influence of menstrual cycle phases on the glycemic control expressed as time in range (% of time between 70-180 mg/dl of interstitial glucose).

SECONDARY OUTCOMES:
Time below range | 1 month
  To assess the influence of menstrual cycle phases on the glycemic control expressed as time in below range (% of time < 70 mg/dl of interstitial glucose).
Time above range | 1 month
  To assess the influence of menstrual cycle phases on time in above range (% of time >180 mg/dl of interstitial glucose).
Caloric intake | 1 month
  To assess the influence of changes in intake throughout the menstrual cycle
Temperature | 1 month
  To collect temperature using a wearable.
Photoplethysmography | 1 month
  To collect photoplethysmography using a wearable.
Accelerometry | 1 month
  To collect acelerometry using a wearable.

CONTACTS AND LOCATIONS:
Overall Officials: Lía Nattero, MD.PhD, Principal Investigator — Diabetes, Obesity and Human Reproduction Research Group (IRYCIS)
Locations (1):
- Lía Nattero-Chávez, Madrid, Madrid, Spain